CLINICAL TRIAL: NCT01637818
Title: Long-term Follow-up of a Randomized Clinical Trial of Lichtenstein's Operation Versus Mesh Plug for Inguinal Hernia Repair
Brief Title: Long-term Follow-up of Lichtenstein's Operation Versus Mesh Plug Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: PD Dr. D. Frey, GZO Wetzikon, Wetzikon, Switzerland (Unknown); Kantonsspital Olten (Other); Prof. J. Metzger, Kantonsspital Luzern, Luzern, Switzerland (Unknown)
Responsible Party: Principal Investigator, Raoul Droeser, MD, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R59
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia repair; long-term follow-up; Surgical technique
MeSH Terms: conditions — Hernia, Inguinal | interventions — Opiate Alkaloids; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lichtenstein's Operation (Other)
  Interventions: Procedure: Lichtenstein's operation; Drug: Opiate; Drug: Paracetamol; Drug: non-steroidal anti-inflammatory drug
- Mesh Plug Repair (Other)
  Interventions: Procedure: Mesh Plug Repair; Drug: Opiate; Drug: Paracetamol; Drug: non-steroidal anti-inflammatory drug

INTERVENTIONS:
Procedure: Lichtenstein's operation
  Arms: Lichtenstein's Operation
Procedure: Mesh Plug Repair
  Arms: Mesh Plug Repair
Drug: Opiate — Postoperative pain therapy
Drug: Paracetamol — Postoperative pain therapy
Drug: non-steroidal anti-inflammatory drug — Postoperative pain therapy

SUMMARY:
Long-term follow-up of a randomized clinical trial of Lichtenstein's operation versus mesh plug for inguinal hernia repair based on the following published study "Randomized clinical trial of Lichtenstein's operation versus mesh plug for inguinal hernia repair. Br J Surg. 2007 Jan;94(1):36-41."

Primary endpoints is recurrence.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older, patients who became 40 in the year of the operation were included (6 patients younger than 40 years were included because of explicit patient's wish).
* provision of written informed consent,
* symptomatic unilateral or bilateral inguinal hernia.

Exclusion Criteria:

* presence of a femoral hernia,
* history of hernia repair with mesh,
* type I diabetes,
* presence of local or diffuse infection (urine, skin, lung, sepsis),
* immune deficiency,
* severe medical problems contraindicating safe induction of general anaesthesia or elective surgery,
* pregnancy,
* malignant tumours and
* life expectancy of less than 2 years

Min Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 1999-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Recurrence | 6 years
  Recurrence after hernia operation (Lichtenstein's operatin versus mesh plug)

SECONDARY OUTCOMES:
Pain | 6 years
  Pain measurement after inguinal hernia repair by visual analog scale (Lichtenstein's operatin versus mesh plug)
Reoperation | 6 years
  Reoperation after inguinal hernia repair (Lichtenstein's operatin versus mesh plug)
Sensitivity | 6 years
  Sensitivity after inguinal hernia repair (Lichtenstein's operatin versus mesh plug: 0 = normal, 1 = reduced, 2 = neuralgia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Frey, MD, Principal Investigator — GZO Wetzikon; Markus Zuber, Prof., Principal Investigator — Kantonsspital Olten; Jürg Metzger, Prof., Principal Investigator — Luzerner Kantonsspital; Rachel Rosenthal, Prof., Principal Investigator — University Hospital, Basel, Switzerland; Raoul Droeser, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Frey DM, Wildisen A, Hamel CT, Zuber M, Oertli D, Metzger J. Randomized clinical trial of Lichtenstein's operation versus mesh plug for inguinal hernia repair. Br J Surg. 2007 Jan;94(1):36-41. doi: 10.1002/bjs.5580. PMID 17094166
- [Derived] Droeser RA, Dell-Kuster S, Kurmann A, Rosenthal R, Zuber M, Metzger J, Oertli D, Hamel CT, Frey DM. Long-term follow-up of a randomized controlled trial of Lichtenstein's operation versus mesh plug repair for inguinal hernia. Ann Surg. 2014 May;259(5):966-72. doi: 10.1097/SLA.0000000000000297. PMID 24169195